CLINICAL TRIAL: NCT05245591
Title: A Randomized, Controlled, Phase II/III Trial to Evaluate the Efficacy and Safety of U101 Oral Capsules in Radiation-induced Cystitis
Brief Title: Radiation Cystitis Treated With Pentosan Polysulfate Sodium Trial
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: TCM Biotech International Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202108161MIPD
Record Dates: First submitted 2022-01-23; First posted 2022-02-18 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-01

CONDITIONS: Radiation Cystitis
MeSH Terms: interventions — Pentosan Sulfuric Polyester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pentosan Polysulfate Sodium (Experimental): U101 is available as a capsule containing 100 milligrams (mg) of pentosan polysulfate sodium. Subjects will be administered U101 at a dose of 300 milligrams (mg) three times daily (tid) for the initial 8 weeks and then 200 milligrams (mg) twice daily (bid) for another 8 weeks during the study.
  Interventions: Drug: Pentosan Polysulfate Sodium 100 MG Oral Capsule
- Placebo Control (Placebo Comparator): Placebo to match U101 is available as a capsule in 100 milligrams (mg). Subjects will be administered placebo at a dose of 300 milligrams (mg) three times daily (tid) for the initial 8 weeks and then 200 milligrams (mg) twice daily (bid) for another 8 weeks during the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentosan Polysulfate Sodium 100 MG Oral Capsule — Pentosan Polysulfate Sodium 100 mg three times daily (tid) for 0-8 weeks Pentosan Polysulfate Sodium 100 mg twice daily (bid) for 9-16 weeks
  Other Names: Urosan; ELMIRON; PPS
  Arms: Pentosan Polysulfate Sodium
Drug: Placebo — Placebo 100 mg three times daily (tid) for 0-8 weeks Placebo 100 mg twice daily (bid) for 9-16 weeks
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pentosan polysulfate sodium versus placebo and in patients with radiation cystitis who have received radiation therapy in pelvic region.

DETAILED DESCRIPTION:
RCT-PPS is a phase II/III study evaluating the efficacy, safety, and tolerability of pentosan polysulfate sodium (PPS) versus placebo to patients with radiation cystitis who have received radiation therapy in pelvic region.

Approximately 72 patients were planned to be randomized in RCT-PPS trial in a 1:1 ratio to treatment with either PPS or placebo. Patients will receive oral treatment with 16 weeks (PPS 100mg three times a day for 8 weeks and then with PPS 100mg twice daily for another 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in the study protocol.
2. Patients must be ≥20 years of age
3. Patients must have received definitive radiation therapy for cancer in pelvic area.
4. Time from the end of radiation therapy to radiation cystitis must be longer than 6 months.
5. Radiation cystitis with lower urinary tract symptoms or hematuria.

Exclusion Criteria:

1. Abnormal liver function with indication of AST, ALT, or total bilirubin ≥ 1.5 times higher than normal
2. Abnormal renal function with serum creatinine ≥ 1.5 times higher than normal
3. Abnormal coagulation profile with PT/INR higher than normal
4. Thrombocytopenia with platelet counts < 100,000/μL
5. Pregnant or breastfeeding, expecting to pregnancy, or positive for pregnancy test
6. Patients who have systemic inflammatory symptoms during screening period (ie, fever up to 38℃ or WBC counts >12,000/μL)
7. Patients with known urinary tract infection within 6 months of randomization.
8. Any previous intravesical instillation within 6 months of randomization (ie, hyaluronic acid instillation)
9. Any previous hyperbaric oxygen therapy within 6 months of randomization
10. Any previous treatment with pentosan polysulfate sodium within 6 months of randomization
11. Has history of thrombocytopenia, hemophilia or bladder cancer
12. Has known history of Human Immunodeficiency Virus (HIV) or organ transplantation
13. Has known history of drug allergy to pentosan polysulfate sodium
14. Has hematuria caused by clinically active urolithiasis or urothelial carcinoma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complete remission in lower urinary tract symptoms and hematuria | From date of randomization throughout the treatment period up to 5 years
  Number of participants without lower urinary tract symptoms and hematuria assessed by ESOU 2019 and CTCAE v5.0
Time to complete remission | From date of randomization to study completion up to 5 years
  Time from randomization to complete remission of lower urinary tract syndromes and hematuria
Time to hematuria recurrence | From date of randomization to study completion up to 5 years
  Time from randomization to recurrence of hematuria
Assessment of quality of life | From date of randomization to study completion up to 5 years
  Functional Assessment of 36-Item Short Form Survey (SF-36)
Assessment of symptoms | From date of randomization to study completion up to 5 years
  Functional Assessment of Expanded Prostate Cancer Index Composite-26 (EPIC-26)

SECONDARY OUTCOMES:
Duration of hospitalization | From date of randomization to study completion up to 5 years
  Overall days of hospitalization due to radiation cystitis
Number of invasive procedures | From date of randomization to study completion up to 5 years
  Percentage of patients underwent transurethral cauterization of bladder bleeders or transurethral clots evacuation.
Number of adverse events | From date of randomization to study completion up to 5 years
  Percentage of patients with any adverse event (AE), adverse event (AE) leading to study drug discontinuation, serious adverse event (SAE), and adverse event (AE) related to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Yuan Huang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No